CLINICAL TRIAL: NCT03906877
Title: Early UVFP Management Based on Neurological Evidences UVFP = Unilateral Vocal Fold Paralysis
Brief Title: Early UVFP Management Based on Neurological Evidences (UVFP = Unilateral Vocal Fold Paralysis)
Acronym: IONS-UVFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/03OCT/365
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Unilateral Vocal Cord Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Injection laryngoplasty group (IL) (Experimental): The patients in the first group will receive an IL of hyaluronic acid in the paralyzed vocal fold within a maximum of three months after the onset of symptoms. The Ear-Noise-Throat (ENT) physician will perform the injection in office, under topical anaesthesia.
  Interventions: Procedure: Acid hyaluronic injection laryngoplasty; Other: Sham of voice therapy
- Voice therapy group (VT) (Experimental): Patients from the second group will be involved in 15 sessions of thirty minutes of voice therapy, twice a week, and will have to do home practice. Patients will have to record these training sessions. Initiation of this intervention should also take place within the first three months after the onset of symptoms. They will also receive an injection of physiological saline under the skin of the neck (sham of injection).
  Interventions: Behavioral: Voice therapy; Other: Sham of injection
- Sham group (Sham Comparator): The patients of the third group will be treated following the traditional wait-and-see policy. They will receive an injection of physiological saline under the skin of the neck and will be seen during 15 sessions of 30 minutes, twice a week. Therefore, this will be a sham procedure for both IL and VT.
  Interventions: Other: Sham of injection; Other: Sham of voice therapy

INTERVENTIONS:
Procedure: Acid hyaluronic injection laryngoplasty — Hyaluronic acid is injected into the paralyzed vocal fold
  Arms: Injection laryngoplasty group (IL)
Behavioral: Voice therapy — 15 sessions of thirty minutes of voice therapy, twice a week, and home practice.
  This voice management will be specific to unilateral vocal fold paralysis and will focus on three objectives: reinforcement of the vocal muscle, glottal closure and glottal opening. These three objectives will be worked through different vocal exercises (on voiced phonemes) and breathing exercises
  Arms: Voice therapy group (VT)
Other: Sham of injection — Injection of physiological saline under the skin of the neck (sham of injection).
  Arms: Sham group; Voice therapy group (VT)
Other: Sham of voice therapy — 15 sessions of thirty minutes of voice therapy, twice a week, and home practice.
  This voice management will not be specific to UVFP but may allow patients to improve their vocal gesture.
  Arms: Injection laryngoplasty group (IL); Sham group

SUMMARY:
The aim of this study is to understand how early intervention could impact reinnervation of the recurrent laryngeal nerve (which innervates the vocal cord), recovery of mobility of the paralyzed vocal cord and / or vocal recovery in the case of unilateral vocal fold paralysis. To achieve this goal we must therefore carry out a complete outcomes assessment of different intervention methods (voice therapy and injection laryngoplasty), which are offered to UVFP (unilateral vocal fold paralysis) patients in the early stage (< 3 months). Their respective impacts on the central and peripheral nervous system and on the voice quality will be assessed, taking into account factors related to the severity of the paralysis.

ELIGIBILITY:
Inclusion Criteria:

- Unilateral paralysis in abduction of the vocal cords may be included in the study.

Exclusion Criteria:

* Wear a pacemaker or other implanted devices (prostheses ...).
* Wear metal clips, metal in the head, or an adjustable brain drain.
* Wear non-removable dental appliances (except fillings).
* Wear cardiac valve prostheses.
* Have worked the metals.
* Have a tattoo containing metal particles.
* Have implanted jewelry (e.g., piercing).
* Being prone to epileptic seizures.
* Take medications that alter cortical excitability.
* Have had a brain surgery.
* Suffer from intracranial hypertension.
* Be pregnant or breastfeeding recently.
* Present allergies that are incompatible with the experimental protocol.
* Have an abnormal hearing loss in view of their age, identified with tonal and / or vocal audiometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Laryngeal recurrent nerve reinnervation | 9 to 12 months after paralysis
  Defined through qualitative laryngeal electromyography
Recovery of the vocal fold mobility | 9 to 12 months after paralysis
  Videostroboscopy examination to analyse vocal folds movements in three dimensions
Voice recovery | 9 to 12 months after paralysis
  Multidimensional voice assessment (based on anamnestic interview, Maximum Phonation Time in sec, Mean Air Flow in ml/sec, Mean subglottic pressure in cmH2O, Jitter in %, Shimmer in %, Noise-to-harmonic ratio, phonetogram, smoothed cepstral peak prominence in %, Voice Handicap Index - VHI-30 (*total* : 0-120, higher value = worse outcome), Medical Outcomes Study 36-item Short Form Healthy Survey (*8 subscales* : 0-100, higher value = better outcome, Eating Assessment Tool-10 (*total*: 0-40, higher value = worse outcome), GRBAS-I (*6 subscales* : 0-3, higher value = worse outcome), Acoustic Voice Quality Index, Dysphonia Severity Index (DSI = 0.13 x MPT + 0.0053 x F(0)-High - 0.26 x I-Low - 1.18 x Jitter (%) + 12.4),Tonal and vocal audiometries in dB)
Changes in the neuronal pathways involved in the processing of the proprioceptive and auditory inputs | 9 to 12 months after paralysis
  Functional magnetic resonance imaging examination (tomodensitometry and connectivity)
Central auditory processes | Within 3 months after paralysis
  Auditory perception tasks performed using an audio headset

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Desuter, Principal Investigator — SSS/MEDE and SSS/IONS/NEUR
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No